CLINICAL TRIAL: NCT03788187
Title: Role of Persistant Organics Pollutants in the Metastatic Potential of Malignant Breast Tumor.
Brief Title: Persistant Organics Pollutants in Breast Cancer.
Acronym: METAPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Georges Pompidou Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); ONIRIS (Industry)
Responsible Party: Principal Investigator, Koual Meriem, Associate professor, European Georges Pompidou Hospital
Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2013-A00663-42
Record Dates: First submitted 2018-12-03; First posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer; Persistant Organic Pollutants; Lymph Node Metastases
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Analyzing the concentrations of 46 POPs in both adipose tissue and serum samples from breast tumor patients (benign, malignant with and without lymph node metastasis).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood test sample
Other: Peritumoral adipose tissue sample

SUMMARY:
Persistant Organics Pollutants (POP) accumulate in the adipose tissue (AT) and could modulate tumor progression as part of the microenvironment. The investigators tested the hypothesis that POPs exposure may be associated with breast cancer metastasis analyzing the concentrations of 46 POPs in both adipose tissue and serum samples from breast tumor patients (benign, malignant with and without lymph node metastasis)

DETAILED DESCRIPTION:
The investigators set up a longitudinal prospective monocentric cohort study in the gynecologic-oncologic surgery department of European Hospital Georges-Pompidou, with patients undergoing partial or total mastectomies, lymph node biopsies or axillary lymph node removal and sampling of the adipocytic tumour microenvironment to measure POPs using gas chromatography coupled to high-resolution mass spectrometry. The objective is to analyze the concentrations of 46 POPs including polychlorinated dibenzo(p)dioxins and furans (PCDD/Fs), polychlorinated biphenyls (PCBs), polybromodiphenyl ethers (PBDEs) and polybromobiphenyls (PBBs) in both adipose tissue (AT) and serum samples from breast tumor patients (benign, malignant with and without lymph node metastasis).

ELIGIBILITY:
Inclusion Criteria:

* Patient with breast tumor: benign or malignant
* Tumor size at least 1cm or palpable tumor
* Undergoing a breast surgery in European Georges Pompidou hospital
* Understanding the protocol and who signed a written consent

Exclusion Criteria: patients unable to give informed consent

* Dementia
* Guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2013-12-27 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Metastatic lymph node status based of persistant organic pollutants level measured by by gas chromatography coupled to high-resolution mass spectrometry. | Sampling the day of surgery
  Correlation between 1) the concentrations of 46 persistant organic pollutants (including polychlorinated dibenzo(p)dioxin and furan, PCBs, polybromodiphenyl ethers and polybromobiphenyls measured by by gas chromatography coupled to high-resolution mass spectrometry on double sector instruments (JEOL MS 700D and 800D) after electron impact ionization (70 eV), operating at 10000 resolutions (10% valley) and in the single ion monitoring (SIM) acquisition mode) in both adipose tissue and serum samples and 2) breast cancer status (with and without lymph node metastasis)

SECONDARY OUTCOMES:
Pro metastatic genes messenger ribonucleic acid (mARN) expression in the tumor based of metastatic lymph node status and persistant pollutants level. | 2 years
  Correlation between the mRNA levels of metastatic biomarkers measured by quantitative reverse transcriptase polymerase chain reaction amplification (PCR) in tumors (based of metastatic lymph node status) and the levels of persistant organic pollutants measured by gas chromatography coupled to high-resolution mass spectrometry.
  List of genes measured : Epithelial-to-mesenchymal (ECadherin, SNAIL, SLUG), matrix metalloproteases, metabolism, vascular endothelial grown factor, stem-cell properties, hormon receptor, inflammatory genes, xenobiotic receptor Aryl Hydrocarbon receptor (AhR).

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie BATS, MD, PhD, Principal Investigator — European Hospital Georges Pompidou